CLINICAL TRIAL: NCT01225211
Title: A Phase 2, Multicenter, Double-Blinded, Placebo-Controlled, Multiple-Dose Study to Evaluate Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Lumacaftor Monotherapy, and Lumacaftor and Ivacaftor Combination Therapy in Subjects With Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: Study of VX-809 Alone and in Combination With VX-770 in Cystic Fibrosis (CF) Patients Homozygous or Heterozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: VX09-809-102; 2010-020413-90 (EudraCT Number)
Record Dates: First submitted 2010-10-15; First posted 2010-10-20 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Cohort 1: Placebo (Placebo Comparator): Participants homozygous (HO) for the F508del-CF transmembrane conductance regulator gene (CFTR) mutation received lumacaftor matched placebo once daily (qd) (Day 1 through Day 14), followed by lumacaftor matched placebo qd in combination with ivacaftor matched placebo every 12 hours (q12h) (Day 15 through Day 21).
  Interventions: Drug: Lumacaftor Placebo; Drug: Ivacaftor Placebo
- Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h (Experimental): Participants homozygous for the F508del-CFTR mutation received 200 milligram (mg) of lumacaftor (LUM) qd (Day 1 through Day 14), followed by 200 mg of lumacaftor qd in combination with 150 mg of ivacaftor (IVA) q12h (Day 15 through Day 21).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (Experimental): Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor alone qd (Day 1 through Day 14), followed by 200 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 15 through Day 21).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 2 and 3: Placebo (HO and HE) (Placebo Comparator): Participants homozygous or heterozygous for the F508del-CFTR mutation received lumacaftor matched placebo qd (Day 1 through Day 28), followed by lumacaftor matched placebo in combination with ivacaftor matched placebo q12h (Day 29 through Day 56).
  Interventions: Drug: Lumacaftor Placebo; Drug: Ivacaftor Placebo
- Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO) (Experimental): Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor alone qd (Day 1 through Day 28), followed by 200 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO) (Experimental): Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor alone qd (Day 1 through Day 28), followed by 400 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO&HE) (Experimental): Participants homozygous or heterozygous for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28), followed by 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO) (Experimental): Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor alone q12h (Day 1 through Day 28), followed by 400 mg of lumacaftor q12h in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor
- Cohort 4: Placebo (Placebo Comparator): Participants heterozygous for the F508del-CFTR mutation received lumacaftor matched placebo in combination with ivacaftor matched placebo q12h (Day 1 through Day 56).
  Interventions: Drug: Lumacaftor Placebo; Drug: Ivacaftor Placebo
- Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h (Experimental): Participants heterozygous for the F508del-CFTR mutation received 400 mg of lumacaftor q12h in combination with 250 mg of ivacaftor q12h (Day 1 through Day 56).
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Lumacaftor — Tablet
  Other Names: VX-809, LUM
  Arms: Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h; Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h; Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO); Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO); Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO&HE); Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO); Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Drug: Ivacaftor — Tablet.
  Other Names: VX-770, IVA
  Arms: Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h; Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h; Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO); Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO); Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO&HE); Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO); Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Drug: Lumacaftor Placebo — Matching placebo tablet.
  Arms: Cohort 1: Placebo; Cohort 2 and 3: Placebo (HO and HE); Cohort 4: Placebo
Drug: Ivacaftor Placebo — Matching placebo tablet.
  Arms: Cohort 1: Placebo; Cohort 2 and 3: Placebo (HO and HE); Cohort 4: Placebo

SUMMARY:
The purpose of this study is to evaluate of the safety, efficacy, pharmacokinetics (PK) and pharmacodynamic (PD) effects of lumacaftor (VX-809) alone and when coadministered with ivacaftor (VX-770) in participants with cystic fibrosis, homozygous or heterozygous for the F508del-CFTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with confirmed diagnosis of CF
* Must have the F508del-CFTR mutation on at least 1 allele.
* FEV1 greater than equal (>=) 40% of predicted normal for age, gender, and height (Knudson standards)(Cohort 1, 2, and 3); FEV1 40-90% of predicted normal for age, gender, and height (Hankinson standards (Cohort 4)
* Participant of child-bearing potential and who are sexually active must meet the contraception requirements

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the participant (e.g., cirrhosis with portal hypertension).
* An acute illness including acute upper or lower respiratory infection, pulmonary exacerbation or changes in therapy (including antibiotics) for pulmonary disease within 14 days (Cohort 1, 2, and 3) or 28 days (Cohort 4) before receiving the first dose of study drug.
* History of solid organ or hematological transplantation.
* History of alcohol abuse or drug addiction in the past year, including cannabis, cocaine, and opiates.
* Ongoing participation in another therapeutic clinical study, or prior participation in an investigational drug study without appropriate washout
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception
* Participants enrolled in Cohort 1 or Cohort 2 will not be eligible for Cohort 3
* Ongoing or prior participation in an investigational drug study within 30 days of the Screening Visit
* Heterozygous participants who participated in Cohort 2 and meet the eligibility criteria for Cohort 4 may participate in Cohort 4
* Evidence of lens opacity or cataract as determined by the ophthalmologic examination (Cohort 4 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (38):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - La Jolla, California
  - Long Beach, California
  - Palo Alto, California
  - Sacramento, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
- Australia (6):
  - Adelaide
  - Brisbane
  - Chermside
  - Nedlands
  - Parkville Victoria
  - Westmead
- Leuven, Belgium
- France (2):
  - Pierre-Bénite, Rhone
  - Paris
- Germany (5):
  - Jena, Thuringia
  - Berlin
  - Bochum
  - Cologne
  - Essen
- New Zealand (2):
  - Auckland
  - Christchurch
- London, United Kingdom

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Rowe SM, McColley SA, Rietschel E, Li X, Bell SC, Konstan MW, Marigowda G, Waltz D, Boyle MP; VX09-809-102 Study Group. Lumacaftor/Ivacaftor Treatment of Patients with Cystic Fibrosis Heterozygous for F508del-CFTR. Ann Am Thorac Soc. 2017 Feb;14(2):213-219. doi: 10.1513/AnnalsATS.201609-689OC. PMID 27898234
- [Derived] Boyle MP, Bell SC, Konstan MW, McColley SA, Rowe SM, Rietschel E, Huang X, Waltz D, Patel NR, Rodman D; VX09-809-102 study group. A CFTR corrector (lumacaftor) and a CFTR potentiator (ivacaftor) for treatment of patients with cystic fibrosis who have a phe508del CFTR mutation: a phase 2 randomised controlled trial. Lancet Respir Med. 2014 Jul;2(7):527-38. doi: 10.1016/S2213-2600(14)70132-8. Epub 2014 Jun 24. PMID 24973281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in each cohort are mutually exclusive. A total of 312 participants were randomized of which one participant did not receive any treatment and a total of 311 participants were treated.
Pre-assignment Details: Study included 4 cohorts which were studied in sequential manner. For results reporting, combined placebo arm was reported for Cohort 2 and 3 and results for these 2 cohorts are reported collectively.
Groups:
- Cohort 4: Placebo: Participants heterozygous for the F508del-CFTR mutation received lumacaftor in combination with ivacaftor matched placebo q12h (Day 1 through Day 56).
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h | Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h | Cohort 2 and 3: Placebo (HO and HE) | Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO&HE) | Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO) | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Started | 21 | 20 | 21 | 27 | 23 | 21 | 42 | 11 | 63 | 62
Completed | 21 | 20 | 20 | 27 | 23 | 21 | 41 | 11 | 62 | 57
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) for Cohort 1, 2, and 3 included all randomized participants who received at least 1 dose of study drug and FAS for Cohort 4 included all randomized participants who received any amount of study drug.
Groups:
- Cohort 1: Placebo: Participants homozygous for the F508del-CFTR mutation received lumacaftor matched placebo qd (Day 1 through Day 14), followed by lumacaftor matched placebo qd in combination with ivacaftor matched placebo q12h (Day 15 through Day 21).
- Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor alone qd (Day 1 through Day 14), followed by 200 mg of lumacaftor qd in combination with 150 mg of ivacaftor q12h (Day 15 through Day 21).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 150 mg q12h | Cohort 1: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h | Cohort 2 and 3: Placebo (HO and HE) | Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO&HE) | Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO) | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h | Total
Number analyzed (Participants) | 21 | 20 | 21 | 27 | 23 | 21 | 42 | 11 | 63 | 62 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 21 | 27 | 23 | 21 | 42 | 11 | 63 | 62 | 311
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 13 | 9 | 11 | 9 | 19 | 5 | 31 | 29 | 144
  Male | 11 | 12 | 8 | 18 | 12 | 12 | 23 | 6 | 32 | 33 | 167

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Safety and Tolerability Based on Adverse Events (AEs)
Description: AE: any untoward medical occurrence in a participant during study; irrespective of relationship with treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after informed consent. AE includes serious AEs (SAEs) as well as Non-SAEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Number of participants with AEs and SAEs are reported. AE that started at/after initial dosing of study drug, or increased in severity after initial dosing of study drug is considered treatment-emergent. Results are reported separately for monotherapy period (Period 1: Day 1 to Day 14) and combination therapy period (Period 2: Day 15 to Day 21).
Time Frame: Cohort 1: Day 1 up to 28 days after last dose (Last dose = Day 21)
Population: Cohort 1 Safety Set included all participants who received at least 1 dose of study drug in Cohort 1. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- Cohort 1: Placebo - Period 1: Participants homozygous for the F508del-CFTR mutation received lumacaftor matched placebo qd (Day 1 through Day 14).
- Cohort 1: LUM 200 mg qd - Period 1: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor alone qd (Day 1 through Day 14).
- Cohort 1: Placebo - Period 2: Participants homozygous for the F508del-CFTR mutation received lumacaftor matched placebo qd in combination with ivacaftor matched placebo q12h (Day 15 through Day 21).
- Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor qd in combination with 150 mg of ivacaftor q12h (Day 15 through Day 21).
- Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 15 through Day 21).
Arm/Group | Cohort 1: Placebo - Period 1 | Cohort 1: LUM 200 mg qd - Period 1 | Cohort 1: Placebo - Period 2 | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2
Number analyzed (Participants) | 21 | 41 | 21 | 20 | 20
participants
  Participants with any AEs | 12 | 29 | 15 | 14 | 12
  Participants with SAEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Cohort 2 and 3: Safety and Tolerability Based on Adverse Events (AEs)
Description: Detailed description is provided in Outcome Measure 1. Results are reported separately for monotherapy period (Period 1: Day 1 to Day 28) and combination therapy period (Period 2: Day 29 to Day 56).
Time Frame: Cohort 2 and 3: Day 1 up to 28 days after last dose (Last dose = Day 56)
Population: Cohort 2 and 3 Safety Set included all participants who received at least 1 dose of study drug in Cohort 2 or 3. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- Cohort 2 and 3: Placebo (HO and HE) - Period 1: Participants homozygous or heterozygous for the F508del-CFTR mutation received lumacaftor matched placebo qd (Day 1 through Day 28).
- Cohort 2: LUM 200 mg qd - Period 1: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor alone qd (Day 1 through Day 28).
- Cohort 2: LUM 400 mg qd - Period 1: Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor alone qd (Day 1 through Day 28).
- Cohort 2: LUM 600 mg qd - Period 1: Participants homozygous or heterozygous for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28).
- Cohort 3: LUM 400 mg q12h - Period 1: Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor alone q12h (Day 1 through Day 28).
- Cohort 2 and 3: Placebo (HO and HE) - Period 2: Participants homozygous or heterozygous for the F508del-CFTR mutation received lumacaftor matched placebo in combination with ivacaftor matched placebo q12h (Day 29 through Day 56).
- Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2: Participants homozygous for the F508del-CFTR mutation received 200 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
- Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2: Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
- Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO&HE) - Period 2: Participants homozygous or heterozygous for the F508del-CFTR mutation received 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
- Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2: Participants homozygous for the F508del-CFTR mutation received 400 mg of lumacaftor q12h in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
Arm/Group | Cohort 2 and 3: Placebo (HO and HE) - Period 1 | Cohort 2: LUM 200 mg qd - Period 1 | Cohort 2: LUM 400 mg qd - Period 1 | Cohort 2: LUM 600 mg qd - Period 1 | Cohort 3: LUM 400 mg q12h - Period 1 | Cohort 2 and 3: Placebo (HO and HE) - Period 2 | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO&HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2
Number analyzed (Participants) | 27 | 23 | 21 | 42 | 11 | 27 | 21 | 20 | 38 | 11
participants
  Participants with any AEs | 23 | 18 | 18 | 37 | 7 | 20 | 12 | 15 | 26 | 10
  Participants with SAEs | 1 | 2 | 0 | 3 | 2 | 4 | 0 | 1 | 4 | 1

3. Primary Outcome: Cohort 4: Safety and Tolerability Assessed by Number of Participants With AEs and SAEs
Description: AEs and SAEs are defined in Outcome Measure 1.
Time Frame: Cohort 4: Day 1 up to 28 days after last dose (Last dose = Day 56)
Population: Cohort 4 Safety Set included all participants who received at least 1 dose of study drug in Cohort 4.
Measure: Number; unit: participants
Groups:
- Cohort 4: Active Study Drug: Participants heterozygous for the F508del-CFTR mutation received 400 mg of lumacaftor q12h in combination with 250 mg of ivacaftor q12h (Day 1 through Day 56).
Arm/Group | Cohort 4: Placebo | Cohort 4: Active Study Drug
Number analyzed (Participants) | 63 | 62
participants
  Participants with any AEs | 53 | 52
  Participants with SAEs | 5 | 9

4. Primary Outcome: Cohort 1: Absolute Change From Day 14 in Sweat Chloride at Day 21
Time Frame: Cohort 1: Day 14, Day 21
Population: Cohort 1 Full Analysis Set included all randomized participants who received at least 1 dose of study drug in Cohort 1. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 | Cohort 1: Placebo - Period 2
Number analyzed (Participants) | 19 | 14 | 17
millimole per liter (mmol/L) | -2.131 [-5.381 to 1.119] | -9.128 [-12.893 to -5.362] | 0.548 [-2.955 to 4.052]
Statistical Analysis 1: Comparison: Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 vs Cohort 1: Placebo - Period 2; Test type: Superiority or Other; p = 0.267, ANCOVA; LS Mean difference = -2.679, 95% CI 2-sided [-7.484 to 2.125]
Statistical Analysis 2: Comparison: Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 vs Cohort 1: Placebo - Period 2; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean difference = -9.676, 95% CI 2-sided [-14.801 to -4.551]

5. Primary Outcome: Cohort 2 And 3: Absolute Change From Day 28 in Sweat Chloride at Day 56
Time Frame: Cohort 2 and 3: Day 28, Day 56
Population: Cohort 2 and 3 Full Analysis Set included all randomized participants who received at least 1 dose of study drug in Cohort 2 or 3. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2: Participants homozygous for the F508del-CFTR mutation received 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
- Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2: Participants heterozygous for the F508del-CFTR mutation received 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
Arm/Group | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 | Cohort 2 and 3: Placebo (HO and HE) - Period 2
Number analyzed (Participants) | 21 | 19 | 20 | 17 | 9 | 24
mmol/L | 0.321 [-4.208 to 4.849] | -1.043 [-5.800 to 3.714] | -2.900 [-7.542 to 1.743] | -1.240 [-6.287 to 3.807] | -2.154 [-9.177 to 4.870] | 1.627 [-2.661 to 5.915]
Statistical Analysis 1: Comparison: Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 vs Cohort 2 and 3: Placebo (HO and HE) - Period 2; Test type: Superiority or Other; p = 0.680, ANCOVA; LS Mean difference = -1.306, 95% CI 2-sided [-7.565 to 4.953]
Statistical Analysis 2: Comparison: Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 vs Cohort 2 and 3: Placebo (HO and HE) - Period 2; Test type: Superiority or Other; p = 0.409, ANCOVA; LS Mean difference = -2.670, 95% CI 2-sided [-9.053 to 3.712]
Statistical Analysis 3: Comparison: Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2 vs Cohort 2 and 3: Placebo (HO and HE) - Period 2; Test type: Superiority or Other; p = 0.161, ANCOVA; LS Mean difference = -4.526, 95% CI 2-sided [-10.888 to 1.835]
Statistical Analysis 4: Comparison: Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2 vs Cohort 2 and 3: Placebo (HO and HE) - Period 2; Test type: Superiority or Other; p = 0.396, ANCOVA; LS Mean difference = -2.867, 95% CI 2-sided [-9.543 to 3.810]
Statistical Analysis 5: Comparison: Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 vs Cohort 2 and 3: Placebo (HO and HE) - Period 2; Test type: Superiority or Other; p = 0.365, ANCOVA; LS Mean difference = -3.780, 95% CI 2-sided [-12.028 to 4.467]

6. Primary Outcome: Cohort 4: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 56
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. ppFEV1 (predicted for age, gender, and height) was calculated using the Hankinson method.
Time Frame: Cohort 4: Baseline, Day 56
Population: Cohort 4 Full Analysis Set included all randomized participants who received any amount of study drug in Cohort 4. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 60 | 55
percent predicted of FEV1 | -1.23 (0.801) | -0.62 (0.829)
Statistical Analysis 1: Comparison: Cohort 4: Placebo vs Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h; Test type: Superiority or Other; p = 0.5978, Mixed Model Repeated Measure (MMRM); LS Mean difference = 0.60, 95% CI 2-sided [-1.66 to 2.86]

7. Secondary Outcome: Cohort 1: Absolute Change From Baseline in Sweat Chloride at Day 14
Time Frame: Cohort 1: Baseline, Day 14
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Cohort 1: LUM 200 mg qd - Period 1 | Cohort 1: Placebo - Period 1
Number analyzed (Participants) | 36 | 17
mmol/L | -4.442 [-7.141 to -1.742] | -1.668 [-5.606 to 2.271]

8. Secondary Outcome: Cohort 2 And 3: Absolute Change From Baseline in Sweat Chloride at Day 14
Time Frame: Cohort 2: Baseline, Day 14
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Cohort 2: LUM 600 mg qd (HO) - Period 1: Participants homozygous for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28).
- Cohort 2: LUM 600 mg qd (HE) - Period 1: Participants heterozygous for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28).
Arm/Group | Cohort 2: LUM 200 mg qd - Period 1 | Cohort 2: LUM 400 mg qd - Period 1 | Cohort 2: LUM 600 mg qd (HO) - Period 1 | Cohort 2: LUM 600 mg qd (HE) - Period 1 | Cohort 3: LUM 400 mg q12h - Period 1 | Cohort 2 and 3: Placebo (HO and HE) - Period 1
Number analyzed (Participants) | 19 | 17 | 21 | 17 | 11 | 25
mmol/L | -6.490 [-11.226 to -1.755] | -5.901 [-10.910 to -0.892] | -9.442 [-13.953 to -4.931] | -3.137 [-8.167 to 1.893] | -9.179 [-15.470 to -2.888] | 0.048 [-4.162 to 4.258]

9. Secondary Outcome: Cohort 4: Absolute Change From Baseline in Sweat Chloride at Day 56
Time Frame: Cohort 4: Baseline, Day 56
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 59 | 54
mmol/L | -0.78 (1.230) | -11.82 (1.281)

10. Secondary Outcome: Cohort 1: Absolute Change From Day 14 in FEV1 at Day 21
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Cohort 1: Day 14, Day 21
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 | Cohort 1: Placebo - Period 2
Number analyzed (Participants) | 20 | 18 | 21
liters | 0.128 [0.030 to 0.225] | 0.015 [-0.094 to 0.124] | -0.046 [-0.138 to 0.047]

11. Secondary Outcome: Cohort 1: Absolute Change From Day 14 in ppFEV1 at Day 21
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 1: Day 14, Day 21
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 | Cohort 1: Placebo - Period 2
Number analyzed (Participants) | 20 | 18 | 21
percent predicted of FEV1 | 3.46 [0.87 to 6.05] | 0.63 [-2.20 to 3.46] | -1.44 [-3.89 to 1.01]

12. Secondary Outcome: Cohort 2 and 3: Absolute Change From Day 28 in ppFEV1 at Day 56
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 2 and 3: Day 28, Day 56
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 | Cohort 2 and 3: Placebo (HO and HE) - Period 2
Number analyzed (Participants) | 21 | 20 | 20 | 17 | 10 | 27
percent predicted of FEV1 | 1.96 [-0.84 to 4.76] | 1.99 [-0.87 to 4.84] | 6.15 [3.27 to 9.02] | 2.29 [-0.82 to 5.39] | 6.09 [2.02 to 10.16] | -1.57 [-4.24 to 1.09]

13. Secondary Outcome: Cohort 2 and 3: Relative Change From Day 28 in ppFEV1 at Day 56
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 2 and 3: Day 28, Day 56
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 | Cohort 2 and 3: Placebo (HO and HE) - Period 2
Number analyzed (Participants) | 21 | 20 | 20 | 17 | 10 | 24
percent change | 3.13 [-1.29 to 7.54] | 2.98 [-1.52 to 7.48] | 9.70 [5.17 to 14.23] | 4.30 [-0.59 to 9.19] | 8.24 [1.83 to 14.65] | -2.05 [-6.25 to 2.15]

14. Secondary Outcome: Cohort 2 and 3: Absolute Change From Baseline in ppFEV1 at Day 28 and 56
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 2 and 3: Baseline, Day 28 and 56
Population: Cohort 2 and 3 Full Analysis Set included all randomized participants who received at least 1 dose of study drug in Cohort 2 or 3. Here, n = participants evaluable for specified category for each arm, respectively. Number of participants analysed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Groups:
- Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO): Participants homozygous for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28), followed by 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
- Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HE): Participants heterozygous (HE) for the F508del-CFTR mutation received 600 mg of lumacaftor alone qd (Day 1 through Day 28), followed by 600 mg of lumacaftor qd in combination with 250 mg of ivacaftor q12h (Day 29 through Day 56).
Arm/Group | Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HE) | Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO) | Cohort 2 and 3: Placebo (HO and HE)
Number analyzed (Participants) | 23 | 21 | 21 | 21 | 11 | 27
percent predicted of FEV1
  Day 28: (n= 21, 20, 20, 18, 11, 27) | 0.21 [-2.77 to 3.19] | -1.35 [-4.39 to 1.69] | -2.62 [-5.67 to 0.42] | -3.82 [-7.03 to -0.61] | -4.52 [-8.65 to -0.39] | -0.03 [-2.68 to 2.62]
  Day 56: (n= 21, 20, 20, 17, 10, 24) | 1.82 [-1.28 to 4.91] | 0.64 [-2.52 to 3.80] | 3.59 [0.41 to 6.77] | -1.68 [-5.12 to 1.75] | 2.16 [-2.34 to 6.66] | -2.02 [-4.97 to 0.93]

15. Secondary Outcome: Cohort 2 and 3: Relative Change From Baseline in FEV1 at Day 28 and 56
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 2 and 3: Baseline, Day 28 and 56
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort 2: LUM 200 mg qd/LUM 200 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 400 mg qd/LUM 400 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HO) | Cohort 2: LUM 600 mg qd/LUM 600 mg qd+IVA 250 mg q12h (HE) | Cohort 3: LUM 400 mg q12h/LUM 400 mg q12h+IVA 250 mg q12h (HO) | Cohort 2 and 3: Placebo (HO and HE)
Number analyzed (Participants) | 23 | 21 | 21 | 21 | 11 | 27
percent change
  Day 28: (n= 21, 20, 20, 18, 11, 27) | 0.24 [-4.27 to 4.75] | -1.15 [-5.75 to 3.45] | -3.13 [-7.74 to 1.48] | -5.46 [-10.32 to -0.60] | -6.39 [-12.65 to -0.14] | 1.89 [-2.12 to 5.90]
  Day 56: (n= 21, 20, 20, 17, 10, 24) | 2.51 [-2.21 to 7.23] | 1.72 [-3.09 to 6.53] | 5.55 [0.70 to 10.39] | -2.34 [-7.57 to 2.89] | 2.96 [-3.90 to 9.81] | -2.42 [-6.91 to 2.08]

16. Secondary Outcome: Cohort 4: Relative Change From Baseline in Percent Predicted FEV1 at Day 56
Description: FEV1 and ppFEV1 are defined in Outcome Measure 6.
Time Frame: Cohort 4: Baseline, Day 56
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 60 | 55
percent change | -2.20 (1.373) | -0.69 (1.423)

17. Secondary Outcome: Cohort 2 and 3: Absolute Change From Day 28 in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Day 56
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Cohort 2 and 3: Day 28, Day 56
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 | Cohort 2 and 3: Placebo (HO and HE) - Period 2
Number analyzed (Participants) | 21 | 20 | 20 | 17 | 10 | 25
units on a scale | 3.3 [-3.6 to 10.1] | 7.9 [0.8 to 14.9] | 8.9 [1.9 to 15.9] | 5.5 [-2.1 to 13.1] | 11.2 [1.3 to 21.1] | -8.6 [-14.9 to -2.2]

18. Secondary Outcome: Cohort 4: Absolute Change From Baseline in CFQ-R Respiratory Domain Score at Day 56
Description: CFQ-R respiratory domain is defined in Outcome Measure 17.
Time Frame: Cohort 4: Baseline, Day 56
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 60 | 55
units on a scale | -0.82 (1.802) | 5.66 (1.864)

19. Secondary Outcome: Cohort 4: Absolute Change From Baseline in Body Mass Index (BMI) at Day 56
Description: BMI was defined as weight in kilogram (kg) divided by height*height in square meter (m^2).
Time Frame: Cohort 4: Baseline, Day 56
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 60 | 56
kg/m^2 | 0.08 (0.075) | -0.04 (0.077)

20. Secondary Outcome: Cohort 4: Absolute Change From Baseline in Weight at Day 56
Time Frame: Cohort 4: Baseline, Day 56
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Number analyzed (Participants) | 60 | 56
kg | 0.16 (0.211) | -0.11 (0.216)

ADVERSE EVENTS:
Time Frame: Cohort 1: Day 1 up to 28 days after last dose (Last dose = Day 21); Cohort 2 and 3: Day 1 up to 28 days after last dose (Last dose = Day 56); Cohort 4: Day 1 up to 28 days after last dose (Last dose = Day 56)
Arm/Group | Cohort 1: LUM 200 mg qd - Period 1 | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 | Cohort 1: Placebo - Period 1 | Cohort 1: Placebo - Period 2 | Cohort 2: LUM 200 mg qd - Period 1 | Cohort 2: LUM 400 mg qd - Period 1 | Cohort 2: LUM 600 mg qd - Period 1 | Cohort 3: LUM 400 mg q12h - Period 1 | Cohort 2 and 3: Placebo (HO and HE) - Period 1 | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO&HE) - Period 2 | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 | Cohort 2 and 3: Placebo (HO and HE) - Period 2 | Cohort 4: Placebo | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/20 | 0/20 | 0/21 | 0/21 | 2/23 | 0/21 | 3/42 | 2/11 | 1/27 | 0/21 | 1/20 | 4/38 | 1/11 | 4/27 | 5/63 | 9/62
Other Adverse Events (participants affected / at risk) | 29/41 | 14/20 | 12/20 | 12/21 | 15/21 | 17/23 | 18/21 | 37/42 | 6/11 | 23/27 | 12/21 | 15/20 | 26/38 | 10/11 | 20/27 | 53/63 | 51/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: LUM 200 mg qd - Period 1 (N=41) | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 (N=20) | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 (N=20) | Cohort 1: Placebo - Period 1 (N=21) | Cohort 1: Placebo - Period 2 (N=21) | Cohort 2: LUM 200 mg qd - Period 1 (N=23) | Cohort 2: LUM 400 mg qd - Period 1 (N=21) | Cohort 2: LUM 600 mg qd - Period 1 (N=42) | Cohort 3: LUM 400 mg q12h - Period 1 (N=11) | Cohort 2 and 3: Placebo (HO and HE) - Period 1 (N=27) | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 (N=21) | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 (N=20) | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO&HE) - Period 2 (N=38) | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 (N=11) | Cohort 2 and 3: Placebo (HO and HE) - Period 2 (N=27) | Cohort 4: Placebo (N=63) | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h (N=62)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spirometry abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CYSTIC FIBROSIS LUNG (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATION ABNORMAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: LUM 200 mg qd - Period 1 (N=41) | Cohort 1: LUM 200 mg qd+IVA 150 mg q12h - Period 2 (N=20) | Cohort 1: LUM 200 mg qd+IVA 250 mg q12h - Period 2 (N=20) | Cohort 1: Placebo - Period 1 (N=21) | Cohort 1: Placebo - Period 2 (N=21) | Cohort 2: LUM 200 mg qd - Period 1 (N=23) | Cohort 2: LUM 400 mg qd - Period 1 (N=21) | Cohort 2: LUM 600 mg qd - Period 1 (N=42) | Cohort 3: LUM 400 mg q12h - Period 1 (N=11) | Cohort 2 and 3: Placebo (HO and HE) - Period 1 (N=27) | Cohort 2: LUM 200 mg qd+IVA 250 mg q12h (HO) - Period 2 (N=21) | Cohort 2: LUM 400 mg qd+IVA 250 mg q12h (HO) - Period 2 (N=20) | Cohort 2: LUM 600 mg qd+IVA 250 mg q12h (HO&HE) - Period 2 (N=38) | Cohort 3: LUM 400 mg q12h+IVA 250 mg q12h (HO) - Period 2 (N=11) | Cohort 2 and 3: Placebo (HO and HE) - Period 2 (N=27) | Cohort 4: Placebo (N=63) | Cohort 4: LUM 400 mg q12h+IVA 250 mg q12h (N=62)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 8 (8) | 12 (13) | 1 (1) | 6 (6) | 3 (5) | 5 (5) | 5 (6) | 3 (4) | 6 (6) | 12 (15) | 13 (16)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 6 (7) | 2 (2) | 5 (5) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 5 (7)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 4 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 9 (10)
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
RESPIRATION ABNORMAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 7 (8) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 9 (9) | 17 (20)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG HYPERINFLATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 5 (6)
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED VISCOSITY OF BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROLONGED EXPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 7 (10) | 5 (5)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 10 (10)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUNNEL VISION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 4 (5) | 5 (7) | 1 (1) | 4 (4) | 4 (7) | 1 (2) | 5 (9) | 0 (0) | 2 (2) | 7 (10) | 2 (3) | 5 (7) | 11 (18) | 3 (4)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 7 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 7 (10) | 5 (5)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 8 (8) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 7 (9) | 7 (7)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISTAL ILEAL OBSTRUCTION SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
FAECAL VOLUME INCREASED (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIP SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST-TUSSIVE VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STEATORRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 4 (6)
PYREXIA (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 9 (10) | 7 (7)
PAIN (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
APPLICATION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
FEELING HOT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
GLUCOSE URINE PRESENT (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROTHROMBIN TIME PROLONGED (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY FUNCTION TEST DECREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (3)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
BLOOD IMMUNOGLOBULIN E INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD SODIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 3 (4) | 3 (3)
BACTERIAL DISEASE CARRIER (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOAESTHESIA FACIAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH FOLLICULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTIC FIBROSIS LUNG (Congenital, familial and genetic disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 7 (7) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MENSTRUATION DELAYED (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYELID OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 7 (8)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood immunoglobulin G increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interleukin level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIA URINE IDENTIFIED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CULTURE THROAT POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGUS SPUTUM TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEIN URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE KETONE BODY PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPLICATION SITE IRRITATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEDIAL TIBIAL STRESS SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTEBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL RASH (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.